CLINICAL TRIAL: NCT04039997
Title: A Comparison of Two Chest Compression Techniques Among Laypersons. A Prospective, Randomized Simulation Study
Brief Title: How to Learn Cardiopulmonary Resuscitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lazarski University (Other)
Collaborators: Wroclaw Medical University (Other); The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Łukasz Szarpak, Associate Professor, Lazarski University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: CPR_NET
Record Dates: First submitted 2019-07-29; First posted 2019-07-31 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Resuscitation; Chest Compression; Quality
Keywords: cardiopulmonary resuscitation; medical simulation; basic life support; chest compression; feedback device

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chest compression without cpr feedback device (Experimental): teaching resuscitation without application of cpr feedback device
  Interventions: Other: Manual chest compression
- Chest compression with cpr feedback device (Experimental): teaching resuscitation with application of CPRMeter - cpr feedback device
  Interventions: Device: CPRMeter

INTERVENTIONS:
Device: CPRMeter — teaching resuscitation with application of cpr feedback device
  Arms: Chest compression with cpr feedback device
Other: Manual chest compression — Manual chest compression
  Arms: Chest compression without cpr feedback device

SUMMARY:
the aim of the study is to evaluate two methods of teaching cardiopulmonary resuscitation in the context of chest compression quality. We will evaluate the usefulness of the application cpr feedback device (CPRMeter) for quality of chest compression.

ELIGIBILITY:
Inclusion Criteria:

* give voluntary consent to participate in the study
* no medical experience

Exclusion Criteria:

* not meet the above criteria
* wrist or low back diseases
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2019-07-20 (Actual); Primary Completion 2019-08-03 (Actual); Study Completion 2019-08-03 (Actual)

PRIMARY OUTCOMES:
chest compressions effectiveness | 1 day
  the percentage of correct chest compressions relative to the total number of chest compressions

SECONDARY OUTCOMES:
depth | 1 day
  correct depth according to European Resuscitation Council 2015 guidelines for cardiopulmonary resuscitation
pressure point | 1 day
  correct pressure point according to European Resuscitation Council 2015 guidelines for cardiopulmonary resuscitation
Complete pressure release | 1 day
  Complete pressure release measure by manikin software
Rate of chest compression | 1 day
  correct chest compressions rate according to European Resuscitation Council 2015 guidelines for cardiopulmonary resuscitation

CONTACTS AND LOCATIONS:
Overall Officials: Lukasz Szarpak, Study Chair — Lazarski University
Locations (1):
- Lazarski Univerisity, Warsaw, Masovia, Poland

IPD SHARING:
Plan to Share IPD: Undecided
after finish study, we will share data on https://repod.pon.edu.pl/pl/